CLINICAL TRIAL: NCT04084899
Title: The Effect of Continuous Positive Airway Pressure Therapy on Lung Hyperinflation in Patients With Obstructive Sleep Apnoea
Brief Title: The Effect of CPAP on Lung Hyperinflation in Patients With OSA
Status: Completed | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Responsible Party: Principal Investigator, Milan Sova, Principal Investigator, Head of Sleep Laboratory, Department of Respiratory Medicine, University Hospital Olomouc
Other Study IDs: OSAS_bodypletysmo
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Continuous Positive Airway Pressure; Lung hyperinflation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Continuous Positive Airway Pressure: Patient treated with continuous positive airway pressure
  Interventions: Device: Continuous Positive Airway Pressure therapy

INTERVENTIONS:
Device: Continuous Positive Airway Pressure therapy — Standard treatment with continuous positive airway pressure

SUMMARY:
Assessment of the lung hyperinflation by bodypletysmography in patients with obstructive sleep apnoea treated with continuous positive airway pressure therapy.

DETAILED DESCRIPTION:
Rationale:

Obstructive sleep apnoea (OSA) is characterized by repetitive closure of upper airways leading to apnoea (complete airflow cessation) or hypopnoea (airflow limitation > 50% + blood oxygen desaturation > 3% or airflow limitation > 30% blood oxygen desaturation > 4%). The prevalence of lung hyperinflations in sleep apnoea patients and effect of continuous positive airway pressure (CPAP) therapy is not known.

Process:

Subjects included in the study will be obstructive sleep apnoea (OSA) patients diagnosed by respiratory polysomnography performed in the Sleep Laboratory, Department of Respiratory Medicine, University Hospital Olomouc.

Bodypletysmography will be performed in the time of OSA diagnosis and after 3 months of CPAP therapy.

Data will be statistically evaluated after completion of the target number of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnoea syndrome indicated for CPAP therapy (Apnoea- Hypopnoea index ˃ 15)

Exclusion Criteria:

* - Bilevel positive airway pressure therapy
* Total lung capacity < 80% lower limit of normal values
* Obstructive ventilatory disorder
* Change in body weight ˃ 10%
* Change in smoking status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obstructive sleep apnoea syndrome indicated for CPAP therapy
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Change of Vital Capacity (VC) (ml) | 3 months
  Percentage change of Vital Capacity after 3 months of CPAP therapy.
Change of Forced Expiratory Volume in 1 second (FEV1) (ml) | 3 months
  Percentage change of Forced Expiratory Volume in 1 second after 3 months of CPAP therapy.
Change of Total Lung Capacity (TLC) (ml) | 3 months
  Percentage change of Total Lung Capacity after 3 months of CPAP therapy.
Change of Residual Volume (RV) (ml) | 3 months
  Percentage change of Residual Volume after 3 months of CPAP therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Milan Sova, MD, Ph.D., Principal Investigator — Department of Respiratory Medicine, University Hospital Olomouc
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: Undecided